CLINICAL TRIAL: NCT00282087
Title: Adjuvant Treatment of High Risk Uterine Leiomyosarcoma With Gemcitabine/Docetaxel Followed by Doxorubicin: A Phase II Trial
Brief Title: Adjuvant Chemotherapy for High Risk Uterine Leiomyosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC005; MSKCC05-128 (Other: Memorial Sloan-Kettering Cancer Center)
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2014-12-01 (Estimated); Status verified 2014-11

CONDITIONS: Leiomyosarcoma; Uterine Neoplasm
Keywords: early stage; high grade; uterine leiomyosarcoma; adjuvant treatment
MeSH Terms: conditions — Leiomyosarcoma; Uterine Neoplasms | interventions — Gemcitabine; Docetaxel; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- gemcitabine/docetaxel then doxorubicin (Other): Gemcitabine 900 mg/m2 IV over 90 minutes days 1 and 8 Docetaxel 75 mg/m2 IV day 8 (pre-medication dexamethasone 4-8 mg p.o. bid for 3 days, starting 12-24 hours prior to docetaxel). Doxorubicin 60 mg/m2 IVP every 21 days for 4 cycles (recommend use of central venous catheter access).
  Interventions: Drug: gemcitabine, docetaxel, doxorubicin

INTERVENTIONS:
Drug: gemcitabine, docetaxel, doxorubicin — Cycles = 28 days

SUMMARY:
The purpose of this trial is to study the benefits of giving chemotherapy to women after they have had surgical resection of their primary disease and have no evidence of disease remaining(known as adjuvant therapy). The major objective of this study is to determine the progression free survival. The goal is to prevent relapse or recurrence of their uterine leiomyosarcoma.

DETAILED DESCRIPTION:
Patients with a diagnosis of early-stage uterine leiomyosarcoma have a 70% chance of relapse or recurrence of their disease. Patients enrolled in this trial will receive 4 cycles of gemcitabine and docetaxel followed by 4 cycles of adriamycin. Following completion of chemotherapy, they will be have repeat imaging at regular intervals to monitor for disease recurrence along with periodic clinical evaluations.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* high risk uterine LMS, FIGO stage I or II
* pathology review of LMS high grade and /or mitotic rate greater than or equal to 5 mitoses/10 hpf
* no longer than 12 weeks from surgical resection of cancer
* no evidence of residual disease
* ECOG 0 or 1
* ANC ≥ 1,500, hemoglobin ≥ 8.0, platelets ≥100,000
* creatinine ≤ 1.5 x institutional upper limits of normal
* adequate liver function
* neuropathy (sensory and motor) ≤ CTC grade 1
* negative pregnancy test
* signed consent

Exclusion Criteria:

* patients with other invasive malignancies
* prior therapy with gemcitabine or docetaxel or doxorubicin
* hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* women who are breast feeding
* cardiac ejection fraction <50%
* prior pelvic irradiation
* treatment with hormone replacement or anti-hormonal agents or other cytotoxic agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2006-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martee L. Hensley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (12):
- United States (12):
  - Washington Cancer Institute/Washington Hospital Center (Medstar), Washington D.C., District of Columbia
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - Winship Cancer Institute at Emory University, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - St. Vincent Gynecologic Oncology, Indianapolis, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Pennsylvania Oncology Hematology Associates, Philadelphia, Pennsylvania
  - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Hensley ML, Wathen JK, Maki RG, Araujo DM, Sutton G, Priebat DA, George S, Soslow RA, Baker LH. Adjuvant therapy for high-grade, uterus-limited leiomyosarcoma: results of a phase 2 trial (SARC 005). Cancer. 2013 Apr 15;119(8):1555-61. doi: 10.1002/cncr.27942. Epub 2013 Jan 18. PMID 23335221
- See also: SARC Website — http://www.sarctrials.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was multi-center study open at 11 major medical centers across the United States.
Groups:
- Women Treated With Adjuvant Regimen for High Risk Uterine LMS: Gemcitabine 900 mg/m2 on days 1 and 8 intravenously over 90 minutes, followed by Docetaxel 75 mg/m2 on day 8 intravenously over 1 hour.
Period: Overall Study
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Started | 47
Completed | 46 (One patient died during cycle 1 of treatment because of infectious complications of AIDS.)
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 44
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 47

OUTCOME MEASURES:

1. Primary Outcome: Two-year Progression-free Survival Among Women Treated With This Adjuvant Regimen for High Risk Uterine LMS
Time Frame: Every 3 months up to two years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 46
percentage of participants | 78 [67 to 91]
Statistical Analysis 1: Comparison: Women Treated With Adjuvant Regimen for High Risk Uterine LMS; The primary endpoint is progression-free survival time, with progression defined as a patient having evidence of recurrent LMS on follow-up evaluation and CT scan. Futility monitoring will be based on the accumulating right-censored PFS time data. The monitoring rules will be based on a Bayesian model; Test type: Superiority or Other; p = 0.15, Bayesian Posterior Probability; Two year PFS = 78, 95% CI 2-sided [67 to 91]

2. Secondary Outcome: Tolerability/Toxicity of This Regimen
Description: Unacceptable toxicity is defined as grade 3 or 4 non-hematologic toxicity events that are considered to be treatment-related, excluding alopecia and fatigue.
Time Frame: Every 28 days during dosing and then every 3 months thereafter until patient comes off study
Measure: Number; unit: number of major toxicity events
Groups:
- Women Treated With Adjuvant Regimen for High Risk Uterine LMS: Number of major toxicity events
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 46
number of major toxicity events | 6

3. Secondary Outcome: Correlation Between Age and Tumor Response to Treatment (PFS)
Time Frame: 2 years
Measure: Median (Full Range); unit: years
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 47
years | 53 [37 to 70]
Statistical Analysis 1: Comparison: Women Treated With Adjuvant Regimen for High Risk Uterine LMS; Age correlation with progression-free survival for patients on study treatment; Test type: Superiority or Other; Cox Proportional Hazards; Hazard Ratio (HR) = -0.00269

4. Secondary Outcome: Correlation Between Menopausal Status at Diagnosis and Tumor Response to Treatment (PFS)
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 47
participants
  Postmenopausal | 43
  Premenopausal | 4
Statistical Analysis 1: Comparison: Women Treated With Adjuvant Regimen for High Risk Uterine LMS; Menopausal status at diagnosis correlation with progression-free survival for patients on study treatment; Test type: Superiority or Other; Cox Proportional Hazards; Hazard Ratio (HR) = 0.02

5. Secondary Outcome: Correlation Between Uterine Serosal Involvement and Tumor Response to Treatment (PFS)
Description: AJCC Stage I: No serosal involvement AJCC Stage II: No serosal involement AJCC Stage III: Serosal only
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 47
participants
  AJCC Stage I | 0
  AJCC Stage II | 6
  AJCC Stage III | 41
Statistical Analysis 1: Comparison: Women Treated With Adjuvant Regimen for High Risk Uterine LMS; Uterine serosal involvement correlation with progression-free survival for patients on study treatment; Test type: Superiority or Other; Cox Proportional Hazards; Hazard Ratio (HR) = 0.101

6. Secondary Outcome: Correlation Between Mitotic Rate and Tumor Response to Treatment (PFS)
Description: Mitotic rate is measured in mitoses per 10 high-power fields
Time Frame: 2 years
Measure: Median (Full Range); unit: mitoses per 10 high-power fields
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 47
mitoses per 10 high-power fields | 18 [5 to 83]
Statistical Analysis 1: Comparison: Women Treated With Adjuvant Regimen for High Risk Uterine LMS; Mitotic rate correlation with progression-free survival for patients on study treatment; Test type: Superiority or Other; Cox Proportional Hazards; Hazard Ratio (HR) = -0.00676

7. Secondary Outcome: Correlation Between Estrogen Receptor (ER) Status and Tumor Response to Treatment (PFS)
Time Frame: 2 years
Population: Only 38 of the 47 patients were evaluable
Measure: Number; unit: participants
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 38
participants
  Positive Status | 24
  Negative Status | 14
Statistical Analysis 1: Comparison: Women Treated With Adjuvant Regimen for High Risk Uterine LMS; Estrogen receptor (ER) status correlation with progression-free survival for patients on study treatment; Test type: Superiority or Other; Cox Proportional Hazards; Hazard Ratio (HR) = -0.708

8. Secondary Outcome: Correlation Between Progesterone Receptor (PR) Status and Tumor Response to Treatment (PFS)
Time Frame: 2 years
Population: Only 38 of the 47 patients were evaluable
Measure: Number; unit: participants
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 38
participants
  Positive Status | 19
  Negative Status | 19
Statistical Analysis 1: Comparison: Women Treated With Adjuvant Regimen for High Risk Uterine LMS; Progesterone receptor (PR) status correlation with progression-free survival for patients on study treatment; Test type: Superiority or Other; Cox Proportional Hazards; Hazard Ratio (HR) = -0.906

9. Secondary Outcome: Correlation Between 1988 FIGO Stage and Tumor Response to Treatment (PFS)
Description: Stage I: confined to the uterine corpus Stage II: confined to corpus and cervix Stage IIIA: serosa involvement only (disease could involve the uterine serosa, but patients must have had no other evidence of local spread)
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 47
participants
  FIFO Stage I | 38
  FIGO Stage II | 7
  FIGO Stage III | 2
Statistical Analysis 1: Comparison: Women Treated With Adjuvant Regimen for High Risk Uterine LMS; 1988 FIGO Stage correlation with progression-free survival for patients on study treatment; Test type: Superiority or Other; Cox Proportional Hazards; Hazard Ratio (HR) = 0.207

10. Secondary Outcome: Correlation Between Estrogen Receptor (ER) or Progesterone Receptor (PR) Positive and Tumor Response to Treatment (PFS)
Time Frame: 2 years
Measure: Number; unit: participants
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Number analyzed (Participants) | 47
participants
  ER or PR Positive | 33
  ER and PR Negative | 14
Statistical Analysis 1: Comparison: Women Treated With Adjuvant Regimen for High Risk Uterine LMS; Estrogen receptor (ER) or progesterone receptor (PR) positive correlation with progression-free survival for patients on study treatment; Test type: Superiority or Other; Cox Proportional Hazards; Hazard Ratio (HR) = -0.564

ADVERSE EVENTS:
Arm/Group | Women Treated With Adjuvant Regimen for High Risk Uterine LMS
Serious Adverse Events (participants affected / at risk) | 9/47
Other Adverse Events (participants affected / at risk) | 14/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Women Treated With Adjuvant Regimen for High Risk Uterine LMS (N=47)
Perforation of bowel (Gastrointestinal disorders) | 1 (1)
Hernia (Injury, poisoning and procedural complications) | 1 (1)
Colostomy Reversal (Gastrointestinal disorders) | 1 (1)
Chest Pain (Cardiac disorders) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Neutrophils (Investigations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Throat Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bilirubin (Investigations) | 1 (1)
Platelets (Investigations) | 1 (1)
Fever (General disorders) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Blood clot (Blood and lymphatic system disorders) | 1 (1)
Renal insufficiency (Blood and lymphatic system disorders) | 1 (1)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Women Treated With Adjuvant Regimen for High Risk Uterine LMS (N=47)
myelosuppression (Endocrine disorders) | 14
Hypersensitivity (Immune system disorders) | 10
neuropathy (Nervous system disorders) | 3
Edema (Skin and subcutaneous tissue disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No